CLINICAL TRIAL: NCT01357252
Title: A Multicenter, Double-blind, Randomized, Parallel-group Study to Compare the Effect of 24 Weeks Treatment With Vildagliptin 50mg qd to Placebo as add-on Therapy to Glimepiride in Patients With Type 2 Diabetes Inadequately Controlled With Sulfonylurea Monotherapy.
Brief Title: Vildagliptin add-on to Glimepiride Versus Placebo Added to Glimepiride in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23154
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vildagliptin
  Arms: vildagliptin
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of vildagliptin 50mg qd as add-on therapy to sulfonylurea in patients with type 2 diabetes inadequately controlled with prior sulfonylurea monotherapy as compared to placebo. This study is aimed at supporting the regulatory approval in China of vildagliptin as combination therapy with sulfonylureas in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of T2DM by standard criteria
2. Patients who have received a stable dose of SU for at least 12 weeks prior to Visit 1
3. HbA1c ≥7.5% to ≤ 11.0% at Visit 1 and Visit 3 (Week -1)
4. Age: ≥18 to ≤ 80 years at Visit 1.
5. BMI ≥ 20 and ≤ 40 kg/m^2 at visit 1.

Exclusion Criteria:

1. FPG ≥ 270mg/dl (15.0 mmol/L) at Visit 1 or Visit 3 (Week -1)
2. Severe or repetitive hypoglycemia, as defined in section 3.1, during the run-in period (between Visit 2 and Visit 4)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Fasting Plasma Glucose | 24 weeks
Safety and tolerability (Frequency of adverse events, serious adverse events, and notable laboratory abnormalities) of add-on therapy with vildagliptin 50 mg qd to glimepiride as compared to pbo | 24 weeks
Responder rates - proportion of subjects reaching predefined HbA1c targets | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- China (12):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Zhenjiang, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

REFERENCES:
- [Derived] Yang W, Xing X, Lv X, Li Y, Ma J, Yuan G, Sun F, Wang W, Woloschak M, Lukashevich V, Kozlovski P, Kothny W; all investigators. Vildagliptin added to sulfonylurea improves glycemic control without hypoglycemia and weight gain in Chinese patients with type 2 diabetes mellitus. J Diabetes. 2015 Mar;7(2):174-81. doi: 10.1111/1753-0407.12169. Epub 2014 Jul 29. PMID 24823599